CLINICAL TRIAL: NCT00487682
Title: Dose-finding Study of ASP2151 in Subjects With Herpes Zoster- A Multicenter, Randomized, Double-blind, Valacyclovir Hydrochloride-controlled, Parallel-group, Comparative Study
Brief Title: Dose-finding Study of ASP2151 in Subjects With Herpes Zoster
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15L-CL-221
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Herpes Zoster
Keywords: Valacyclovir hydrochloride; herpes zoster; ASP2151
MeSH Terms: conditions — Herpes Zoster | interventions — ASP2151; Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): ASP2151 low dose
  Interventions: Drug: ASP2151
- 2 (Experimental): ASP2151 middle dose
  Interventions: Drug: ASP2151
- 3 (Experimental): ASP2151 high dose
  Interventions: Drug: ASP2151
- 4 (Active Comparator): Valacyclovir hydrochloride
  Interventions: Drug: Valacyclovir hydrochloride

INTERVENTIONS:
Drug: ASP2151 — oral
  Arms: 1; 2; 3
Drug: Valacyclovir hydrochloride — oral
  Arms: 4

SUMMARY:
To investigate the efficacy and safety of three different doses of ASP2151, as compared to valacyclovir hydrochloride in subjects with herpes zoster, and to determine the recommended clinical dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged from 20 years to under 80 years on the day informed consent is obtained
* Subjects to whom the study drugs can be orally administered within 72 hours after the onset of rash due to herpes zoster
* Subjects in whom protocol-specified observations and assessments are considered possible

Exclusion Criteria:

* Subjects with extremely compromised immune function due to underlying diseases, treatment with Immunosuppressive agents etc., or radiotherapy
* Subjects with a serious underlying disease that corresponds to Grade 3 in the Classification Criteria for teh Seriousness of Adverse Drug Reactions
* Subjects with concurrent malignant tumors, or those with a history of malignant tumors within the past 5 years

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2007-11-13 (Actual); Primary Completion 2008-09-01 (Actual); Study Completion 2008-09-01 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy and safety of ASP2151 with valacyclovir in subjects with Herpes Zoster | 3 months

SECONDARY OUTCOMES:
Improvement of cutaneous symptoms and pain | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Chūbu
  - Hokkaido
  - Kanto
  - Kinki
  - Kyusyu

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial as it meets one or more of the exceptions described on www.clinicalstudydatarequest.com under "Sponsor Specific Details for Astellas."

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=232